CLINICAL TRIAL: NCT00928707
Title: Phase II Study of the Histone-deacetylase Inhibitor GIVINOSTAT (ITF2357) in Combination With Hydroxyurea in Patients With JAK2V617F Positive Polycythemia Vera Non-responder to Hydroxyurea Monotherapy.
Brief Title: Phase II Study of GIVINOSTAT (ITF2357) in Combination With Hydroxyurea in Polycythemia Vera
Acronym: PV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Italfarmaco (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DSC/08/2357/38
Record Dates: First submitted 2009-06-25; First posted 2009-06-26 (Estimated); Results first posted 2019-10-31 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Polycythemia Vera
Keywords: Polycythemia Vera; GIVINOSTAT; ITF2357
MeSH Terms: conditions — Polycythemia Vera | interventions — givinostat; givinostat hydrochloride; Hydroxyurea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GIVINOSTAT + MTD Hydroxyurea (HU)_1 (Experimental): 50 mg o.d. of GIVINOSTAT + maximum tolerated dose (MTD) of Hydroxyurea (HU) monotherapy
  Interventions: Drug: GIVINOSTAT (ITF2357) 50 mg o.d. + MTD Hydroxyurea
- GIVINOSTAT + MTD Hydroxyurea (HU)_2 (Experimental): 50 mg b.i.d. of GIVINOSTAT + maximum tolerated dose (MTD) of Hydroxyurea (HU) monotherapy
  Interventions: Drug: GIVINOSTAT (ITF2357) 50 mg b.i.d. + MTD Hydroxyurea

INTERVENTIONS:
Drug: GIVINOSTAT (ITF2357) 50 mg o.d. + MTD Hydroxyurea — 50 mg o.d. of GIVINOSTAT + MTD of HU monotherapy
  Other Names: GIVINOSTAT (ITF2357); ONCOCARBIDE (HYDROXYUREA)
  Arms: GIVINOSTAT + MTD Hydroxyurea (HU)_1
Drug: GIVINOSTAT (ITF2357) 50 mg b.i.d. + MTD Hydroxyurea — 50 mg b.i.d. of GIVINOSTAT + MTD HU monotherapy
  Other Names: GIVINOSTAT (ITF2357); ONCOCARBIDE (HYDROXYUREA)
  Arms: GIVINOSTAT + MTD Hydroxyurea (HU)_2

SUMMARY:
The primary objective of the study was to evaluate the efficacy of Givinostat in combination with hydroxyurea in patients with JAK2V617F-positive Polycythemia Vera (PV) non-responders to the maximum tolerated dose of hydroxyurea monotherapy.

The secondary objectives of this study were:

* To evaluate the safety and tolerability of Givinostat in combination with hydroxyurea in patients with JAK2V617Fpositive PV non-responders to the maximum tolerated dose of hydroxyurea monotherapy;
* To explore the impact in terms of efficacy and tolerability of Givinostat 50 mg dose escalation in patients not achieving at least a partial response at the time when the primary endpoint was assessed (week 12);
* To evaluate the molecular response (JAK2 mutated allele burden) by quantitative Real Time-Polymerase Chain Reaction (RT-PCR);
* To evaluate the reduction of the fraction of JAK2V617F positive clonogenic progenitors.

DETAILED DESCRIPTION:
This is a multicentre, randomized, open-label, phase II study testing GIVINOSTAT (ITF2357) in combination with hydroxyurea in a population of patients with JAK2V617F positive Polycythemia Vera non-responders to the maximum tolerated dose of hydroxyurea monotherapy for at least 3 months.

Recruited patients will be randomly assigned to one of the following treatment groups:

* group A: 50 mg o.d. of oral GIVINOSTAT (ITF2357) in combination with the maximum tolerated dose of hydroxyurea monotherapy already in use before admission to the study;
* group B: 50 mg b.i.d. of oral GIVINOSTAT (ITF2357) in combination with the maximum tolerated dose of hydroxyurea monotherapy already in use before admission to the study.

The two groups will be balanced for number and for Centre in order to provide valuable information on both treatment regimens.

In both groups assigned doses shall remain stable until week 12, which is when the primary endpoint is assessed, unless specific tolerability issues arise which impose dose reduction.

After the primary endpoint assessment at week 12, one of the following treatment schedules will be chosen case by case on the basis of the achieved clinical response and continued for up to 12 further weeks:

* Partial or Complete Response at week 12:
* group A: continue 50 mg o.d.;
* group B: continue 50 mg b.i.d.;
* No Response at week 12:
* group A: increase to 50 mg b.i.d.;
* group B: increase to 50 mg t.i.d.. At any time during study course, if toxicity is observed, GIVINOSTAT (ITF2357) treatment will be discontinued until recovery and then restarted at a reduced dose level. The drug will be definitively withdrawn in case of reappearance of toxicity even at a reduced daily dose. Overall, the treatment will last up to a maximum of 24 cumulative weeks of drug administration.

The study will recruit subjects of both genders with an established diagnosis of JAK2V617F positive Polycythemia Vera according to the revised WHO criteria, in need of cytoreductive therapy, non-responders to the maximum tolerated dose of hydroxyurea monotherapy for at least 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Written Informed Consent.
* Age ≥18 years.
* Confirmed diagnosis of Polycythemia Vera according to the revised World Health Organization (WHO) criteria.
* JAK2V617F positivity.
* Non-response to the maximum tolerated dose of hydroxyurea monotherapy for at least 3 months.
* ECOG (Eastern Cooperative Oncology Group) performance status <3.
* Use of an effective means of contraception for women of childbearing potential and men with partners of childbearing potential.
* Willingness and capability to comply with the requirements of the study.

Exclusion Criteria:

* Active bacterial or mycotic infection requiring antimicrobial treatment.
* Pregnancy or lactation.
* A marked baseline prolongation of QT/QTc (corrected) interval (e.g. repeated demonstration of a QTc interval > 450 ms, according to Bazett's correction formula).
* Use of concomitant medications that prolong the QT/QTc interval.
* Clinically significant cardiovascular disease including:

  * Uncontrolled hypertension, myocardial infarction, unstable angin, within 6 months from study start;
  * New York Heart Association (NYHA) Grade II or greater congestive heart failure;
  * History of any cardiac arrhythmia requiring medication (irrespective of its severity);
  * A history of additional risk factors for torsade de pointes (TdP) (e.g., heart failure, hypokalemia, family history of Long QT Syndrome).
* Positive blood test for HIV (Human Immunodeficiency Virus)
* Active HBV (Hepatitis B Virus) and/or HCV (Hepatitis C Virus) infection.
* Platelets count <100x109/L within 14 days before enrolment.
* Absolute neutrophil count <1.2x109/L within 14 days before enrolment.
* Serum creatinine >2xULN (upper limit of normal).
* Total serum bilirubin >1.5xULN.
* Serum aspartate aminotransferase (AST) / alanine aminotransferase (ALT) > 3xULN.
* History of other diseases, metabolic dysfunctions, physical examination findings, or clinical laboratory findings giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug or that might affect interpretation of the results of the study or render the subject at high risk from treatment complications.
* Interferon alpha within 14 days before enrolment.
* Anagrelide within 7 days before enrolment.
* Any other investigational drug within 28 days before enrolment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2009-06; Primary Completion 2011-07 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Rambaldi, MD, Principal Investigator — Azienda Ospedaliera Ospedali Riuniti di Bergamo
Locations (22):
- Italy (22):
  - Azienda Ospedaliero-Universitaria Policlinico Consorziale di Bari, Bari, BA
  - Azienda Ospedaliera Santa Croce e Carle di Cuneo, Cuneo, CN
  - Azienda Ospedaliera di Rilievo Nazionale e di Alta Specializzazione Garibaldi di Catania, Catania, CT
  - Fondazione I. R. C. C. S. - Casa sollievo della sofferenza di San Giovanni Rotondo, San Giovanni Rotondo, FG
  - Azienda Ospedaliero-Universitaria Careggi di Firenze, Florence, FI
  - Azienda Ospedaliera San Gerardo di Monza, Monza, MB
  - Azienda Ospedaliera Universitaria Policlinico "Gaetano Martino" di Messina, Messina, ME
  - Azienda Ospedaliera Ospedali Riuniti "Villa Sofia - Cervello" di Palermo, Palermo, PA
  - Azienda Unità Sanitaria Locale di Pescara, Presidio Ospedaliero "Spirito Santo", Pescara, PE
  - Azienda Ospedaliera Santa Maria della Misericordia di Perugia, Perugia, PG
  - Azienda Ospedaliera Universitaria Pisana, Pisa, PI
  - Azienda Ospedaliera Ospedale San Carlo di Potenza, Potenza, Point
  - Fondazione I.R.C.C.S.-Policlinico San Matteo, Pavia, Pavia, PV
  - Azienda Ospedaliera "Bianchi-Melacrino-Morelli", Reggio Calabria, RC
  - Azienda Ospedaliera Universitaria S. Luigi Gonzaga di Orbassano, Orbassano, TO
  - Azienda Ospedaliero-Universitaria San Giovanni Battista("Le Molinette") di Torino, Torino, TO
  - Ospedale Mauriziano Umberto I, Torino, TO
  - Ospedale San Bortolo di Vicenza, Vicenza, VI
  - Azienda Ospedaliera Ospedali Riuniti di Bergamo, Bergamo
  - Azienda Ospedaliera Universitaria Università degli Studi di Napoli Federico II, Napoli
  - Università "Campus Bio-Medico", Rome, Rome
  - Policlinico Universitario Agostino Gemelli di Roma, Rome

RESULTS

PARTICIPANT FLOW:
Groups:
- GIVINOSTAT +Maximum Tolerated Dose (MTD) of Hydroxyurea (HU)_1: 50 mg o.d. of GIVINOSTAT + maximum tolerated dose (MTD) of hydroxyurea (HU) monotherapy
  GIVINOSTAT (ITF2357) 50 mg o.d. + maximum tolerated dose (MTD) of Hydroxyurea (HU): 50 mg o.d. of GIVINOSTAT + maximum tolerated dose (MTD) of Hydroxyurea (HU) monotherapy
- GIVINOSTAT +Maximum Tolerated Dose (MTD) of Hydroxyurea (HU)_2: 50 mg b.i.d. of GIVINOSTAT + maximum tolerated dose (MTD) of Hydroxyurea (HU) monotherapy
  GIVINOSTAT (ITF2357) 50 mg b.i.d. + maximum tolerated dose (MTD) of Hydroxyurea (HU): 50 mg b.i.d. of GIVINOSTAT + maximum tolerated dose (MTD) of Hydroxyurea (HU) monotherapy
Period: Overall Study
Arm/Group | GIVINOSTAT +Maximum Tolerated Dose (MTD) of Hydroxyurea (HU)_1 | GIVINOSTAT +Maximum Tolerated Dose (MTD) of Hydroxyurea (HU)_2
Started | 23 | 22
Completed | 22 | 22
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety/Intention-to-treat (ITT) population, which included all randomized subjects who received at least one dose of study medication.
Groups:
- GIVINOSTAT + MTD Hydroxyurea_1: 50 mg o.d. of GIVINOSTAT + MTD of HU monotherapy
  GIVINOSTAT (ITF2357) 50 mg o.d. + MTD Hydroxyurea: 50 mg o.d. of GIVINOSTAT + MTD of HU monotherapy
- GIVINOSTAT + MTD Hydroxyurea_2: 50 mg b.i.d. of GIVINOSTAT + MTD of HU monotherapy
  GIVINOSTAT (ITF2357) 50 mg b.i.d. + MTD Hydroxyurea: 50 mg b.i.d. of GIVINOSTAT + MTD HU monotherapy
- Total: Total of all reporting groups
Arm/Group | GIVINOSTAT + MTD Hydroxyurea_1 | GIVINOSTAT + MTD Hydroxyurea_2 | Total
Number analyzed (Participants) | 23 | 22 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 11 | 21
  >=65 years | 13 | 11 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 14 | 15 | 29
Region of Enrollment [Number; unit: participants]
  Italy | 23 | 22 | 45

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Overall Haematological Response at Week 12.
Description: The percentage of patients with overall (complete or partial) response at week 12 were assessed. · Complete response: 1. HCT (Hematocrit) < 45% without phlebotomy, and 2. platelets ≤ 400 x109/L, and 3. WBC (white blood cell) ≤ 10 x 109/L, and 4. no splenomegaly, and 5. no disease related systemic symptoms (microvascular disturbances, pruritus, headache); · Partial response: 1. HCT < 45% without phlebotomy, or 2. fulfilment of at least 3 of the other above mentioned criteria; · No response: any response that did not satisfy the criteria set for partial response.
Time Frame: At week 12 of treatment
Population: Safety/ITT population: included all randomized subjects who received at least one dose of study medication.
Measure: Number (95% Confidence Interval); unit: percentage of particpants
Arm/Group | GIVINOSTAT + MTD Hydroxyurea_1 | GIVINOSTAT + MTD Hydroxyurea_2
Number analyzed (Participants) | 22 | 22
percentage of particpants
  Responder | 54.5 [33.7 to 75.4] | 50.0 [29.1 to 70.9]
  Non responder | 45.5 [24.6 to 66.3] | 50.0 [29.1 to 70.9]

2. Secondary Outcome: Percentage of Patients With Overall Haematological Response at Week 24 by Dose Escalation After Week 12.
Description: Haematological response after a 50 mg increase of the initial Givinostat dose in non-responder patients at the time when the primary endpoint was assessed (week 12).
  * Complete response:
    1. HCT< 45% without phlebotomy, and
    2. platelets ≤ 400 x109/L, and
    3. WBC ≤ 10 x 109/L, and
    4. no splenomegaly, and
    5. no disease related systemic symptoms (microvascular disturbances, pruritus, headache);
  * Partial response:
    1. HCT < 45% without phlebotomy, or
    2. fulfilment of at least 3 of the other above mentioned criteria;
  * No response:
  any response that did not satisfy the criteria set for partial response.
Time Frame: At week 24 of treatment
Population: Safety/Intention to treat (ITT) population included all randomized subjects who received at least one dose of study medication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GIVINOSTAT + MTD Hydroxyurea_1 | GIVINOSTAT + MTD Hydroxyurea_2
Number analyzed (Participants) | 22 | 22
percentage of participants
  Responder | 63.6 [43.5 to 83.7] | 40.9 [20.4 to 61.5]
  Non responder | 36.4 [16.3 to 56.5] | 59.1 [38.5 to 79.6]

3. Secondary Outcome: Change From Baseline of the JAK2V617F Allele Burden by Quantitative RT-PCR
Description: To determine JAK2V617F mutational status, a quantitative RT-PCR (Real Time-Polymerase Chain Reaction) is executed on peripheral blood granulocyte and haematopoietic colonies (with and without hepatocyte growth factors - HGFs).
Time Frame: At weeks 12, 24, at "drop out visit" and at "End of Study" (EOS). EOS stays for 7 days after last drug intake if patient is withdrawn from the study before week 24.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | GIVINOSTAT + MTD Hydroxyurea_1 | GIVINOSTAT + MTD Hydroxyurea_2
Number analyzed (Participants) | 22 | 21
percent change
  Week 12 | -2.6 (8.2) | 0.00 (6.0)
  Week 24 | -3.8 (11.5) | 4.6 (5.7)
  Drop-out | -4.0 (0.00) | -9.5 (20.5)
  EOS | -3.8 (11.1) | 3.0 (8.6)

4. Secondary Outcome: Percentage of Patients With a Reduction of the Fraction of JAK2V617F Positive Clonogenic Progenitor by Timepoints
Description: JAK2V617F genotyping and quantification were performed on gradient-separated mononuclear cells during the pre-treatment evaluations (baseline), halfway through the study (12th weeks) and at the end of the study period (24th weeks).
  Baseline: n=22 (50 mg od); 22 (50 mg bid) Week 12: n=20 (50 mg od); 19 (50 mg bid) Week 24: n=18 (50 mg od); 18 (50 mg bid)
Time Frame: Baseline, at weeks 12 and 24
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | GIVINOSTAT + MTD Hydroxyurea_1 | GIVINOSTAT + MTD Hydroxyurea_2
Number analyzed (Participants) | 22 | 22
percentage of participants
  Baseline - heterozygous | 27.3 | 22.7
  Baseline - homozygous | 72.7 | 72.7
  Baseline - not done | 0 | 4.5
  week 12 - heterozygous: number analyzed (Participants) | 20 | 19
  week 12 - heterozygous | 25.0 | 31.6
  week 12 - homozygous: number analyzed (Participants) | 20 | 19
  week 12 - homozygous | 70.0 | 63.2
  week 12 - not done: number analyzed (Participants) | 20 | 19
  week 12 - not done | 5.0 | 5.3
  week 24 - heterozygous: number analyzed (Participants) | 18 | 18
  week 24 - heterozygous | 22.2 | 11.1
  week 24 - homozygous: number analyzed (Participants) | 18 | 18
  week 24 - homozygous | 72.2 | 77.8
  week 24 - not done: number analyzed (Participants) | 18 | 18
  week 24 - not done | 5.6 | 11.1

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were recorded at weeks 1 ,3, 6, 9, 12, 16, 20 or end of treatment visit (week 24 or 7 days after last drug intake)
Arm/Group | GIVINOSTAT + MTD Hydroxyurea_1 | GIVINOSTAT + MTD Hydroxyurea_2
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 2/22 | 1/22
Other Adverse Events (participants affected / at risk) | 21/22 | 21/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GIVINOSTAT + MTD Hydroxyurea_1 (N=22) | GIVINOSTAT + MTD Hydroxyurea_2 (N=22)
Appendicectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pregnancy of partner (Social circumstances) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GIVINOSTAT + MTD Hydroxyurea_1 (N=22) | GIVINOSTAT + MTD Hydroxyurea_2 (N=22)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 1 (2) | 0 (0)
Curetting of chalazion (Surgical and medical procedures) | 1 (1) | 0 (0)
Asthenia (General disorders) | 2 (2) | 2 (2)
Fatigue (General disorders) | 2 (2) | 1 (1)
Oedema (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (3) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (2) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 3 (3) | 2 (6)
Blood magnesium increased (Investigations) | 2 (2) | 0 (0)
Blood tryglicerides increased (Investigations) | 0 (0) | 1 (4)
Blood urea increased (Investigations) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 2 (2)
Platelet count increased (Investigations) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (3)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (3)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (5) | 7 (8)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 10 (12) | 7 (10)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 2 (3) | 1 (1)
Tongue haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (3) | 1 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Genitourinary tract infection (Infections and infestations) | 0 (0) | 1 (2)
Influenza (Infections and infestations) | 3 (3) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Urogenital infection fungal (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No